CLINICAL TRIAL: NCT00747448
Title: CryoSpray Ablation (TM) GI Patient Registry
Status: Completed | Type: Observational
Sponsor: CSA Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 17-00030
Record Dates: First submitted 2008-09-04; First posted 2008-09-05 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-02

CONDITIONS: Barrett's Esophagus; Esophageal Cancer
Keywords: Barrett's Esophagus; High Grade Dysplasia; Low Grade Dysplasia; Squamous Dysplasia; Esophageal Cancer; CryoSpray Ablation; Cryotherapy; Cryospray
MeSH Terms: conditions — Barrett Esophagus; Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to create a patient registry to collect and analyze post-510K approval information on subjects treated endoscopically with the CryoSpray Ablation™ System.

DETAILED DESCRIPTION:
The proposed registry is a prospective, multi-center study of patients that are being currently undergoing CryoSpray Ablation™. It will also be used to catalogue retrospective data from records of patients already treated with the device. A maximum of 40 investigational sites will participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* The study population consists of patients who are being treated, or were treated, with the CryoSpray Ablation™ System for malignant or pre-malignant conditions of the esophagus, including:

  * Barrett's esophagus with or without dysplasia
  * Squamous dysplasia of the esophagus
  * Esophageal cancer, any stage

Exclusion Criteria:

* Subjects with esophageal lesions whose pathology was not one of the above.
* Subjects with one of the above conditions who were not treated with the CryoSpray Ablation™ System.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients who are being treated, or were treated, with the CryoSpray Ablation™ System for malignant or pre-malignant conditions of the esophagus, including:
  1. Barrett's esophagus with or without dysplasia
  2. Squamous dysplasia of the esophagus
  3. Esophageal cancer, any stage, as evidenced by histology.
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2009-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Primary objectives of the study are to enable analysis of patient outcomes 2 years after final treatment and report on the effectiveness of the device in eradicating, decreasing or downgrading of the lesions. | 2 years post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ann Murphy Legg, RN, Study Director — CSA Medical, Inc.
Locations (6):
- United States (6):
  - The Scripps Research Institute, La Jolla, California
  - University of Maryland Medical Center, Baltimore, Maryland
  - Syosset Hospital, Lake Success, New York
  - University of North Carolina-Chapel Hill, Chapel Hill, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Rhode Island Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johnston MH, Eastone JA, Horwhat JD, Cartledge J, Mathews JS, Foggy JR. Cryoablation of Barrett's esophagus: a pilot study. Gastrointest Endosc. 2005 Dec;62(6):842-8. doi: 10.1016/j.gie.2005.05.008. PMID 16301023
- [Background] Johnston CM, Schoenfeld LP, Mysore JV, Dubois A. Endoscopic spray cryotherapy: a new technique for mucosal ablation in the esophagus. Gastrointest Endosc. 1999 Jul;50(1):86-92. doi: 10.1016/s0016-5107(99)70352-4. PMID 10385730
- [Background] Ell C, May A, Gossner L, Pech O, Gunter E, Mayer G, Henrich R, Vieth M, Muller H, Seitz G, Stolte M. Endoscopic mucosal resection of early cancer and high-grade dysplasia in Barrett's esophagus. Gastroenterology. 2000 Apr;118(4):670-7. doi: 10.1016/s0016-5085(00)70136-3. PMID 10734018
- [Background] Champion G, Richter JE, Vaezi MF, Singh S, Alexander R. Duodenogastroesophageal reflux: relationship to pH and importance in Barrett's esophagus. Gastroenterology. 1994 Sep;107(3):747-54. doi: 10.1016/0016-5085(94)90123-6. PMID 8076761
- [Background] Eisen GM, Sandler RS, Murray S, Gottfried M. The relationship between gastroesophageal reflux disease and its complications with Barrett's esophagus. Am J Gastroenterol. 1997 Jan;92(1):27-31. PMID 8995932
- [Background] Johnston MH. Cryotherapy and other newer techniques. Gastrointest Endosc Clin N Am. 2003 Jul;13(3):491-504. doi: 10.1016/s1052-5157(03)00044-8. PMID 14629105
- [Background] Cash BD, Johnston LR, Johnston MH. Cryospray ablation (CSA) in the palliative treatment of squamous cell carcinoma of the esophagus. World J Surg Oncol. 2007 Mar 16;5:34. doi: 10.1186/1477-7819-5-34. PMID 17367523
- [Background] Pinsonneault C, Fortier J, Donati F. Tracheal resection and reconstruction. Can J Anaesth. 1999 May;46(5 Pt 1):439-55. doi: 10.1007/BF03012943. PMID 10349923